CLINICAL TRIAL: NCT07051603
Title: A Phase 1, Randomized, Double-Blind Placebo-Controlled Single and Multiple Dose Study Plus Food Effect Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of SAL0140 in Healthy Chinese Subjects
Brief Title: SAL0140 Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in a Healthy Chinese Population
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAL0140A101
Record Dates: First submitted 2025-06-17; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Uncontrolled Hypertension
Keywords: SAL0140; Uncontrolled hypertension; Pharmacokinetic; Pharmacodynamic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Doses (SAD, Part A) (Experimental): In this part, 5 ascending dose cohorts (8 participants per cohort) will be studied. Within each cohort, participants will be randomized in a 6:2 ratio to receive either SAL0140 or placebo.
  Interventions: Drug: SAL0140; Drug: SAL0140 placebo
- Experimental: Foode Effect (FE, Part B) (Experimental): 12 participants and single dose food effect cohort. This part is open-label, two sequence, two-period, crossover design. Participants will be randomly assigned to 1 of the 2 crossover sequence
  Interventions: Drug: SAL0140
- Experimental: Single Ascending Doses (MAD, Part C) (Experimental): In this part, 3 ascending dose cohorts (10 participants per cohort) will be studied. Within each cohort, participants will be randomized in an 8:2 ratio to receive either SAL0140 or placebo.
  Interventions: Drug: SAL0140; Drug: SAL0140 placebo

INTERVENTIONS:
Drug: SAL0140 — In this part, SAL0140 tablets will be administered as a single or multiple oral dose.
Drug: SAL0140 placebo — In this part, SAL0140 placebo tablets will be administered as a single or multiple oral dose.
  Arms: Experimental: Single Ascending Doses (MAD, Part C); Single Ascending Doses (SAD, Part A)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability pharmacokinetics and pharmacodynamics of SAL0140 healthy Chinese population.

DETAILED DESCRIPTION:
This trial contains Part A, Part B and Part C, all enrolling healthy Chinese subjects. Part A is a randomized, double-blind, placebo-controlled, single ascending dose study designed to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single oral dose of SAL0140 tablets in healthy Chinese adult participants. Part B is a randomized, open-label, single-dose, two-period, two-sequence, crossover study designed to evaluate the effect of food on the pharmacokinetic characteristics of SAL0140 tablets in healthy Chinese adult participants. Part C is a randomized, double-blind, placebo-controlled, multiple ascending dose study designed to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple oral doses of SAL0140 tablets in healthy Chinese adult participants.

Part A will be conducted first, and Parts B and C will be initiated when appropriate based on the preliminary data obtained during the study. Each participant can only participate in one dose group in any part of the study after dosing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects has fully understood and voluntarily signed the informed consent form, and is able to comply with the requirements and restrictions listed in the informed consent form;
* Male or female aged 18-65 years (including 18 and 65 years old);
* Male body weight ≥50kg, female body weight ≥45kg and body mass index (BMI) between 19.0 - 26.0 kg/m2 (including 19.0 and 26.0, BMI = weight(kg) / height(cm)2) at screening;
* All examinations (including physical examination, vital signs, laboratory tests, ECG, chest X-ray (anterior and lateral views), etc.) show no abnormalities or minor abnormalities deemed non clinical signiant by the investigator;

Exclusion Criteria:

* Subjects with orthostatic tachycardia or orthostatic hypotension at screening; or those with a history of orthostatic hypotension symptoms (such as dizziness, fatigue, blurred vision, pallor upon standing) or orthostatic tachycardia symptoms (such as dizziness, palpitations, tremors, general weakness, blurred vision, exercise intolerance when standing);
* Subjects have used corticosteroids within 3 months prior to dosing;
* Subjects with personal or family history of long QT syndrome, torsades de pointes, or other complex arrhythmias, or family history of sudden death;
* Subjects with prolonged QTcF interval (>450msec) on ECG;
* Subjects with potassium levels above the upper limit of normal (>ULN) or sodium levels below the lower limit of normal (<LLN) in biochemistry tests;
* Subjects with known allergies to excipients in the study drug or history of severe allergic reactions (including food, drugs, insect bites, etc.);
* Subjects with any disease history or current condition that may affect the safety evaluation or drug disposition of the study participant, including but not limited to central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, immune system, psychiatric conditions, metabolic disorders, gastrointestinal surgery (except appendectomy), etc.;
* Subjects have undergone gastric surgery, vagotomy, bowel resection, or any surgery that may interfere with gastrointestinal motility, pH, or absorption;
* Subjects received live or attenuated vaccines within 4 weeks prior to screening;
* Subjects consume excessive tea, coffee, and/or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) daily, or have consumed these beverages within 48h prior to dosing, or cannot stop consuming during the trial;
* Subjects have taken any prescription drugs, over-the-counter medications, Chinese herbs, or dietary supplements (including vitamins, health foods, etc.) within 14 days prior to dosing;
* Subjects with a history of long-term consumption of xanthine-rich or grapefruit-containing beverages or foods, or who have consumed any xanthine-rich or grapefruit products within 48h prior to dosing;
* Subjects have smoked within 3 months prior to screening, or cannot stop using any tobacco products during the trial;
* Subjects have participated in other clinical trials and taken any investigational drugs within 3 months prior to screening;
* Subjects have donated blood or lost blood ≥400 mL, received blood transfusion or blood products within 3 months prior to screening;
* Subjects have had unprotected sexual intercourse within 2 weeks prior to screening; study participants and their spouses or partners who have pregnancy plans, sperm/egg donation plans during the study period until 1 month after dosing, or do not agree to use at least one of the following acceptable effective contraception methods:

  * Correctly placed intrauterine device;
  * Male/female condom used in combination with topical spermicide (i.e., foam, gel, film, cream, or suppository);
  * Male vasectomy or vas deferens ligation;
  * Female bilateral tubal ligation/bilateral salpingectomy or bilateral tubal occlusion surgery (occlusion surgery verified effective by relevant instruments);
  * Abstinence.
* Pregnant or lactating women, or women of childbearing potential with positive pregnancy screening results;
* Subjects are alcoholic or regular drinkers within 3 months prior to screening, i.e., weekly alcohol consumption exceeding 14 standard units (1 unit = 360 mL beer or 45 mL spirits with 40% alcohol content or 150 mL wine) or positive baseline alcohol breath test, or cannot stop using any alcohol-containing products during the trial;
* Subjects positive drug abuse screening or history of drug abuse or previous use of illicit drugs;
* Subjects tested positive for hepatitis B surface antigen, hepatitis C antibody, syphilis antibody, or human immunodeficiency virus (HIV) antibody; Subjects deemed by the investigator to have poor compliance or other factors that unsuitable for participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The rate of Adverse events | from Day 1 to Day8 or Day23 or Day28
  The rate of Adverse events occur during the whole study
The rate of normality or abnormality of electrocardiogram | from Day 1 to Day8 or Day23 or Day28
  The rate of normality or abnormality of electrocardiogram during the whole study

CONTACTS AND LOCATIONS:
Overall Officials: Chongyuan Xu, Ph.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No